CLINICAL TRIAL: NCT02875912
Title: PROSPECTIVE EVALUATION OF FAMILY CARE RITUALS IN THE ICU AND VALIDATION OF THE END-of-Life ScorING-System (ENDING-S), a Multicenter, Multinational Trial
Brief Title: Prospective Evaluation of Family Care Rituals in the ICU
Acronym: FCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: James M. Cox Foundation (Unknown)
Responsible Party: Principal Investigator, Mitchell Levy, Chief of the Division of Pulmonary, Critical Care and Sleep Medicine Rhode Island Hospital, Brown University, Brown University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 763434-9
Record Dates: First submitted 2016-08-04; First posted 2016-08-23 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Stress Disorders, Post-Traumatic; Depression; Anxiety
Keywords: Family; Care Rituals; End of Life; Discordance of care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Death

STUDY DESIGN:
Intervention Model Description: Prospective before and after intervention evaluation
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Family members are surveyed at enrollment, day 5 (if patient is still in ICU), and 90 days post ICU discharge for symptoms of PTSD, depression, and anxiety as well as for concordance of care at enrollment and ICU day 5. Nursing completes surveys while the patient is in the ICU noting what care rituals, if any, are being performed to establish baseline data
- Family Care Rituals Intervention (Experimental): At enrollment, family members are given a handout/pamphlet outlining the Family Care Rituals. They are informed of the opportunity to perform these rituals, but that they are in no way obligated to do so. The families are then surveyed in the same way as they were during the usual care, with nursing completing the same surveys as well to compare against the baseline data
  Interventions: Behavioral: Family Care Rituals

INTERVENTIONS:
Behavioral: Family Care Rituals — Family members being enrolled are given a pamphlet outlining the Family Care Rituals. They are informed of the opportunity to perform these rituals, but that they are in no way obligated to do so.
  Family members are then surveyed at enrollment, and 90 days post ICU discharge for symptoms of PTSD, as well as depression, and anxiety.
  Family members, day-time nursing, and attending physicians are surveyed for concordance of care at enrollment and ICU day 5.
  Demographic information is also collected on the patient and the family members at enrollment Nursing completes surveys while the patient is in the ICU noting what care rituals, if any, are being performed. Additionally, they are asked to complete a survey indicating their opinion of the impact on the care they deliver
  Arms: Family Care Rituals Intervention

SUMMARY:
This study will evaluate whether or not engaging family members of patients admitted to the ICU in "Family Care Rituals" will reduce stress related symptoms of PTSD, depression and anxiety 90 days after patient death or discharge from the ICU. Family Care Rituals are defined as several domains in which family participation may be of benefit, focusing on the 5 physical senses as well as the personal care of the patient and spirituality of the patient

DETAILED DESCRIPTION:
Over the previous century, the location of where people die has shifted from home to either hospitals or nursing homes, with 20% of patients dying in the ICU. Several deficiencies for End-of-Life (EOL) care provided in the ICU have been identified in literature; most of them are related to communication, decision making, sense of control, spirituality, preparation for death, pain and symptom management. Symptoms of stress, anxiety or depression as well as discordance between the perceptions of care by the health care providers (physicians and nurses) and the family members may all be related to these shortcomings. These symptoms are likely from multiple factors in the ICU that strip the family of the ability to provide any direct care or nurturing for their loved one, as families did when people died at home. Moreover, qualitative studies suggest that families want and value a role as a care provider for their loved ones in the ICU. In a pilot study, the investigators identified several domains in which family participation may be of benefit, focusing on the 5 physical senses, personal care of the patient, and spirituality of the patient and family. These areas were incorporated as Family Care Rituals (FCR) in which family members can participate while their loved one is in the ICU

The investigators are conducting a multi-center, multinational prospective evaluation of FCR with the hypothesis that FCR will primarily reduce symptoms of PTSD, as well as anxiety and depression in the surviving family members at 90 days after death or discharge from the ICU. Additionally, the intervention's effect on concordance of care as measured on day of enrollment and ICU day 5 via a questionnaire administered to the family members, the day-time nurse and the attending physician will be evaluated. ICU utilization, family satisfaction, and validation of the END of live scorING System (ENDING-S) are also being evaluated. To understand what care rituals are being performed at the bedside as well as the impact on bedside nursing care, nursing is also completing daily surveys.

The investigators are planning a study of independent cases and controls with 1 control(s) per case. Prior data indicate that the incidence of PTSD in family members is 33%. To reduce the rate of PTSD for family members in the interventional arm to 17%, 114 experimental subjects and 114 control subjects will need to be enrolled to be able to reject the null hypothesis that the failure rates for experimental and control subjects are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. An uncorrected chi-squared statistic will be used to evaluate this null hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Families of patients admitted to the intensive care unit (ICU) with attending physician predicted ICU mortality of greater than 30%.
* Patients with ICU length of stay greater than 4 days, regardless of mortality, are considered for ENDING-S score

Exclusion Criteria:

* Families of patients with an anticipated ICU length of stay less than 24 hours
* Families of patients admitted to the ICU for palliative/comfort care only
* Families of patients with age less than 18
* Families of patients who are pregnant
* Families of patients who are incarcerated
* Family members who are less than 18
* Family members who are pregnant
* Family members who are incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Symptoms of Post-Traumatic Stress Disorder in family members of intensive care patients | 90 days post patient discharge from ICU
  Symptoms of PTSD are measured by the Impact of Events Scale revised (IES-r). This survey is conducted via phone 90 days after patient discharge.

SECONDARY OUTCOMES:
Symptoms of depression in family members of intensive care patients | 90 days post patient discharge from ICU
  Symptoms of Depression are measured by the Hospital Anxiety and Depression Screen (HADS). These surveys are conducted via phone 90 days after patient discharge
Symptoms of anxiety in family members of intensive care patients | 90 days post patient discharge from the ICU
  Symptoms of Anxiety are measured by the Hospital Anxiety and Depression Screen (HADS). These surveys are via phone 90 days after patient discharge
Family satisfaction with ICU care | 90 days post discharge from ICU
  Measured by the Family Satisfaction in the ICU- 24 (FS-ICU-24) questionnaire via phone communication at 90 days
Congruency of goals of care | Evaluated at enrollment and if patient is still in the ICU on hospital day 5 during active enrollment
  Enrolled family members, day time nurse and attending physician are surveyed on enrollment day (day 0) and day 5 with a questionnaire designed to evaluate comfort with the care plan and identify why, if uncomfortable, they are uncomfortable with the care plan
Validation of the End of Life Scoring System (ENDING-S) | Through study completion, anticipated to be 18 months
  Multicenter prospective validation of ENDING-S. This score produces a number based on the following calculation: [ENDING-S = (7.25 ∙ Days of Mechanical ventilation/ICU Length of stay) + (10.45 ∙ Days of Vasoactive drugs/ICU length of stay) + (3 ∙ Sepsis) + (0.3 ∙ ICU Length of stay)] where "sepsis" is binary yes/no as to whether or not the patient is septic. Will also include evaluation of the addition of multi-parametric variables (such as functional status, spiritual and communicative variables) to the ENDING-S to generate a final score based on in hospital morbidity combined with prehospital comorbidities
ICU length of stay | Through study completion, anticipated to be 18 months
  In an effort to evaluate resources used during study period, ICU length of stay will be collected to ascertain whether or not the intervention reduces length of stay
Use of palliative/spiritual care during ICU stay | Through study completion, anticipated to be 18 months
  In an effort to evaluate resources used during study period, data on whether or not a palliative/spiritual care order was placed will be collected to ascertain whether or not the intervention impacts use of these resources
Location of discharge from ICU | Through study completion, anticipated to be 18 months
  In an effort to understand type of discharge (death, another hospital floor, nursing home, hospice, etc), charts will be reviewed for location of discharge from the ICU to ascertain whether or not the intervention impacted discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell M Levy, MD, Principal Investigator — Brown University
Locations (3):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Brown University, Providence, Rhode Island
- Azienda Ospedaliero-Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carson SS, Cox CE, Wallenstein S, Hanson LC, Danis M, Tulsky JA, Chai E, Nelson JE. Effect of Palliative Care-Led Meetings for Families of Patients With Chronic Critical Illness: A Randomized Clinical Trial. JAMA. 2016 Jul 5;316(1):51-62. doi: 10.1001/jama.2016.8474. Erratum In: JAMA. 2017 May 23;317(20):2134. doi: 10.1001/jama.2017.4298. PMID 27380343
- [Background] Silveira MJ, Kim SY, Langa KM. Advance directives and outcomes of surrogate decision making before death. N Engl J Med. 2010 Apr 1;362(13):1211-8. doi: 10.1056/NEJMsa0907901. PMID 20357283
- [Background] White DB. Strategies to Support Surrogate Decision Makers of Patients With Chronic Critical Illness: The Search Continues. JAMA. 2016 Jul 5;316(1):35-7. doi: 10.1001/jama.2016.8691. No abstract available. PMID 27380340
- [Background] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Background] Curtis JR, Back AL, Ford DW, Downey L, Shannon SE, Doorenbos AZ, Kross EK, Reinke LF, Feemster LC, Edlund B, Arnold RW, O'Connor K, Engelberg RA. Effect of communication skills training for residents and nurse practitioners on quality of communication with patients with serious illness: a randomized trial. JAMA. 2013 Dec 4;310(21):2271-81. doi: 10.1001/jama.2013.282081. PMID 24302090
- [Background] Curtis JR, Treece PD, Nielsen EL, Gold J, Ciechanowski PS, Shannon SE, Khandelwal N, Young JP, Engelberg RA. Randomized Trial of Communication Facilitators to Reduce Family Distress and Intensity of End-of-Life Care. Am J Respir Crit Care Med. 2016 Jan 15;193(2):154-62. doi: 10.1164/rccm.201505-0900OC. PMID 26378963
- [Background] Azoulay E, Chevret S, Leleu G, Pochard F, Barboteu M, Adrie C, Canoui P, Le Gall JR, Schlemmer B. Half the families of intensive care unit patients experience inadequate communication with physicians. Crit Care Med. 2000 Aug;28(8):3044-9. doi: 10.1097/00003246-200008000-00061. PMID 10966293
- [Background] Heyland DK, Rocker GM, O'Callaghan CJ, Dodek PM, Cook DJ. Dying in the ICU: perspectives of family members. Chest. 2003 Jul;124(1):392-7. doi: 10.1378/chest.124.1.392. PMID 12853551
- [Background] Angus DC, Barnato AE, Linde-Zwirble WT, Weissfeld LA, Watson RS, Rickert T, Rubenfeld GD; Robert Wood Johnson Foundation ICU End-Of-Life Peer Group. Use of intensive care at the end of life in the United States: an epidemiologic study. Crit Care Med. 2004 Mar;32(3):638-43. doi: 10.1097/01.ccm.0000114816.62331.08. PMID 15090940
- [Background] Reyniers T, Deliens L, Pasman HR, Morin L, Addington-Hall J, Frova L, Cardenas-Turanzas M, Onwuteaka-Philipsen B, Naylor W, Ruiz-Ramos M, Wilson DM, Loucka M, Csikos A, Rhee YJ, Teno J, Cohen J, Houttekier D. International variation in place of death of older people who died from dementia in 14 European and non-European countries. J Am Med Dir Assoc. 2015 Feb;16(2):165-71. doi: 10.1016/j.jamda.2014.11.003. Epub 2014 Dec 18. PMID 25544001
- [Background] Jones C, Skirrow P, Griffiths RD, Humphris G, Ingleby S, Eddleston J, Waldmann C, Gager M. Post-traumatic stress disorder-related symptoms in relatives of patients following intensive care. Intensive Care Med. 2004 Mar;30(3):456-60. doi: 10.1007/s00134-003-2149-5. Epub 2004 Feb 4. PMID 14767589
- [Background] Fumis RR, Ranzani OT, Martins PS, Schettino G. Emotional disorders in pairs of patients and their family members during and after ICU stay. PLoS One. 2015 Jan 23;10(1):e0115332. doi: 10.1371/journal.pone.0115332. eCollection 2015. PMID 25616059
- [Background] Hartog CS, Schwarzkopf D, Riedemann NC, Pfeifer R, Guenther A, Egerland K, Sprung CL, Hoyer H, Gensichen J, Reinhart K. End-of-life care in the intensive care unit: a patient-based questionnaire of intensive care unit staff perception and relatives' psychological response. Palliat Med. 2015 Apr;29(4):336-45. doi: 10.1177/0269216314560007. Epub 2015 Jan 29. PMID 25634628
- [Background] Engstrom A, Soderberg S. The experiences of partners of critically ill persons in an intensive care unit. Intensive Crit Care Nurs. 2004 Oct;20(5):299-308; quiz 309-10. doi: 10.1016/j.iccn.2004.05.009. PMID 15450619
- [Background] McAdam JL, Arai S, Puntillo KA. Unrecognized contributions of families in the intensive care unit. Intensive Care Med. 2008 Jun;34(6):1097-101. doi: 10.1007/s00134-008-1066-z. Epub 2008 Mar 28. PMID 18369593
- [Background] Teno JM, Clarridge BR, Casey V, Welch LC, Wetle T, Shield R, Mor V. Family perspectives on end-of-life care at the last place of care. JAMA. 2004 Jan 7;291(1):88-93. doi: 10.1001/jama.291.1.88. PMID 14709580
- [Background] Hanson LC, Danis M, Garrett J. What is wrong with end-of-life care? Opinions of bereaved family members. J Am Geriatr Soc. 1997 Nov;45(11):1339-44. doi: 10.1111/j.1532-5415.1997.tb02933.x. PMID 9361659
- [Background] Lilly CM, De Meo DL, Sonna LA, Haley KJ, Massaro AF, Wallace RF, Cody S. An intensive communication intervention for the critically ill. Am J Med. 2000 Oct 15;109(6):469-75. doi: 10.1016/s0002-9343(00)00524-6. PMID 11042236
- [Background] Abbott KH, Sago JG, Breen CM, Abernethy AP, Tulsky JA. Families looking back: one year after discussion of withdrawal or withholding of life-sustaining support. Crit Care Med. 2001 Jan;29(1):197-201. doi: 10.1097/00003246-200101000-00040. PMID 11176185
- [Background] Harvey MA. Evolving toward--but not to--meeting family needs. Crit Care Med. 1998 Feb;26(2):206-7. doi: 10.1097/00003246-199802000-00007. No abstract available. PMID 9468150
- [Background] Lynn J, Teno JM, Phillips RS, Wu AW, Desbiens N, Harrold J, Claessens MT, Wenger N, Kreling B, Connors AF Jr. Perceptions by family members of the dying experience of older and seriously ill patients. SUPPORT Investigators. Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments. Ann Intern Med. 1997 Jan 15;126(2):97-106. doi: 10.7326/0003-4819-126-2-199701150-00001. PMID 9005760
- [Background] Pochard F, Azoulay E, Chevret S, Lemaire F, Hubert P, Canoui P, Grassin M, Zittoun R, le Gall JR, Dhainaut JF, Schlemmer B; French FAMIREA Group. Symptoms of anxiety and depression in family members of intensive care unit patients: ethical hypothesis regarding decision-making capacity. Crit Care Med. 2001 Oct;29(10):1893-7. doi: 10.1097/00003246-200110000-00007. PMID 11588447
- [Background] Piers RD, Azoulay E, Ricou B, Dekeyser Ganz F, Decruyenaere J, Max A, Michalsen A, Maia PA, Owczuk R, Rubulotta F, Depuydt P, Meert AP, Reyners AK, Aquilina A, Bekaert M, Van den Noortgate NJ, Schrauwen WJ, Benoit DD; APPROPRICUS Study Group of the Ethics Section of the ESICM. Perceptions of appropriateness of care among European and Israeli intensive care unit nurses and physicians. JAMA. 2011 Dec 28;306(24):2694-703. doi: 10.1001/jama.2011.1888. PMID 22203538
- [Background] Seferian EG, Afessa B. Adult intensive care unit use at the end of life: a population-based study. Mayo Clin Proc. 2006 Jul;81(7):896-901. doi: 10.4065/81.7.896. PMID 16835969
- [Background] Sprung CL, Woodcock T, Sjokvist P, Ricou B, Bulow HH, Lippert A, Maia P, Cohen S, Baras M, Hovilehto S, Ledoux D, Phelan D, Wennberg E, Schobersberger W. Reasons, considerations, difficulties and documentation of end-of-life decisions in European intensive care units: the ETHICUS Study. Intensive Care Med. 2008 Feb;34(2):271-7. doi: 10.1007/s00134-007-0927-1. Epub 2007 Nov 9. PMID 17992508
- [Background] Villa G, De Gaudio AR, Falsini S, Lanini I, Curtis JR. Development of END-of-Life ScorING-System to identify critically ill patients after initial critical care who are highly likely to die: a pilot study. Minerva Anestesiol. 2015 Dec;81(12):1318-28. Epub 2015 Jan 23. PMID 25616205
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Derived] Villa G, Amass T, Giua R, Lanini I, Chelazzi C, Tofani L, McFadden R, De Gaudio AR, OMahony S, Levy MM, Romagnoli S. Validation of END-of-life ScorING-system to identify the dying patient: a prospective analysis. BMC Anesthesiol. 2020 Mar 9;20(1):63. doi: 10.1186/s12871-020-00979-y. PMID 32164567